CLINICAL TRIAL: NCT05796102
Title: Feasibility Study of PET-MRI as a Platform for Image Guidance and Adaptive Radiation Therapy in Patients With Esophagogastric Cancer
Brief Title: PET-MRI Esophagus Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-5780
Record Dates: First submitted 2022-12-09; First posted 2023-04-03 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Esophagogastric Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-MRI (Experimental): PET-MRI in esophagogastric cancers
  Interventions: Procedure: PET-MRI

INTERVENTIONS:
Procedure: PET-MRI — A PET/MRI scan is a two-in-one test that combines images from a positron emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan. Magnetic Resonance Imaging (MRI) provides better soft tissue contrast compared to conventional computerized tomography (CT), and when combined with PET, can potentially provide better visualization of the tumor shape, size, and position.
  Additional MRI imaging will be completed once during radiation treatment, and once after radiation treatment

SUMMARY:
This is a single arm, single centre, investigator initiated study to investigate the feasibility of using PET-MRI imaging in radiation treatment workflow in up to 15 patients with esophagogastric cancer. PET-MRI imaging will be completed before the start of radiation treatment. MRI imaging will be completed during radiation treatment and after radiation treatment. These images will not be used to plan the radiation treatment and routine clinical care will be provided.

The goal of this study is to gather information that will allow the radiation team to include MRI and PET imaging into the radiation treatment workflow for patients with esophageal cancer receiving radiation therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Diagnosed with locally advanced esophageal cancer being considered for conventional RT >4 weeks
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Contraindication for MRI
* Contraindication for Gadolinium (i.e. inability to lie supine for at least 60 minutes)
* Any patient who is pregnant or breastfeeding
* Pacemaker or implanted defibrillator
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of PET-MRI to visualize and assess impact of RT treatments on esophagogastric tumors | 2 years
  Detection of metastases on DWI and gadolinium enhanced T1-weighted 3D VIBE sequences.

SECONDARY OUTCOMES:
Difference in manual GTV segmentation using PET-MRI | 2 years
  Differences in manual GTV segmentation between standard of care treatment plan and study generated treatment plan using PET-MRI.
Quantification of dosimetric advantages of PET-MRI treatment plan | 2 years
  Comparison of dosimetry properties between the standard of care treatment plan and study generated treatment plan using PET-MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada